CLINICAL TRIAL: NCT06081127
Title: A Randomized Pilot Test of the Breast Cancer Pre-habilitation and Prospective Surveillance to Prevent, Detect, and Optimize Physical and Functional Recovery
Brief Title: Breast Cancer Pre-habilitation and Prospective Surveillance to Prevent, Detect, and Optimize Physical and Function
Acronym: B-PREPed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Ann Marie Flores, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00218105
Record Dates: First submitted 2023-10-04; First posted 2023-10-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients assigned to the intervention arm will receive the intervention named Moving On After Breast Cancer (MOve-ABC).
  Interventions: Other: MOve-ABC
- Enhanced Usual Care (EUC) (Experimental): All patients will receive EUC. However, participants assigned to this arm will have only EUC.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: MOve-ABC — The intervention is called Moving On After Breast Cancer (MOve-ABC) and includes:
  1. Three in-person visits for clinical measurements
  2. Enhanced usual care (EUC)
  3. Pre-hab (Pre-Treatment (PT) evaluation and individualized home therapeutic exercise prescription with safe progressions).
  4. Teach Back (HEP, post-op movement precautions)
  5. Self-management education with reinforcement check-ins via text messaging and phone calls at regular intervals.
  Arms: Intervention
Other: Enhanced Usual Care — All patients will receive EUC. However, half of our sample will have only EUC consisting of
  1. Three in-person visits for clinical measurements
  2. Planned oncology treatment (surgery, chemotherapy, radiation)
  3. Nursing education on surgical site and drain care, post-operative movement precautions, pain management
  4. If needed, laboratory and radiological testing to rule out disorders that interfere with treatment outcomes
  5. Monthly monitoring with Patient-Reported Outcomes Measurement Information System - Physical Function (PROMIS-PF) surveys beginning at baseline with alerts from scores = or < 45 (indicating moderate or severe impairment) for physical therapy referral
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The goal of this research study is to determine the feasibility and potential effects of physical therapy and enhanced patient education delivered before breast cancer treatment. Physical therapy before cancer treatment aims to help with early identification and self-management of physical and functional side effects from cancer treatment. Side effects could be joint pain, muscle weakness, or fatigue that contribute to functional impairment.

The main questions this study aims to answer are:

1. Determine the feasibility (acceptability and suitability) and potential effects of an early intervention called 'Moving On-After Breast Cancer' (MOve-ABC) on physical and functional side effects of cancer compared to enhanced usual care in a large academic medical system to help us refine and adjust the intervention in preparation for a large randomized, double-blinded, controlled trial.
2. Determine whether MOve-ABC also affects patient self-management and provider knowledge and behaviors related to detection and management of physical and functional effects associated with cancer.

Participants will be randomly assigned to either of the two arms of the study which are 'Intervention' and 'Enhanced usual care.'

Participants in the intervention arm will receive:

1. Planned care per their oncology physician team plus: 1.1. Patient education on physical function in breast cancer 1.2. Physical therapy evaluation 1.3. Individualized home exercise prescription 1.4. Education materials in the form of a study booklet, study website, text messaging, and phone calls 1.5. Monthly monitoring of physical and functional survey scores to identify the need for physical therapy and provide referrals as needed

Participants in the enhanced usual care arm will receive:

1. Planned care per their oncology physician team plus 1.2. Monthly monitoring of their physical functional scores to identify the need for physical therapy and provide referrals as needed

All participants will attend three in-person visits for clinical measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed Breast Cancer (BC) (stages 0-4) deemed eligible by the oncology physician team to undergo intent-to-cure treatment
* Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Scale score of 0 (Fully active, able to carry on all pre-disease performance without restriction), 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house- work, office work); or 2 (Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours)
* Patients must be Female [Note: Males are not included as BC in males is less than 1% of all cases]
* Patients must be English speaking
* Patients must be age ≥ 18 years
* Patients must have regular access to a mobile phone that can receive text messages and phone calls
* Patients must have the ability to understand and the willingness to sign a written informed consent document prior to registration on study

Exclusion Criteria:

* Patient with any prior malignancy (except non-melanoma skin)
* Patients with an ECOG Performance Scale score of 3 (Capable of only limited self-care; confined to bed or chair more than 50% of waking hours), 4 (Completely disabled; cannot carry on any self-care; totally confined to bed or chair) or 5 (dead)
* History of pre-existing upper extremity functional impairment, lymphedema, central nervous system damage, other systemic medical condition (e.g. fibromyalgia, rheumatoid arthritis, diabetes)
* Actively receiving physical therapy at the time of recruitment and baseline measurement
* Patients with brain metastasis with adverse events attributable to the metastasis ≥ grade 3
* Patients who are pregnant or lactating
* Patients with any issue that would limit their ability to comply with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Feasibility in terms of percentage of participants completing the study protocol | Through study completion, an average of one year
Number of study participants with a score of less than 45 on the "Patient Reported Outcome Measurement Information System Physical Function Custom Form v2.0 Computerized Patient Reported Outcomes" | Baseline, Month 1, Month 2, Month 3, Month 4, Month 6
  This questionnaire is a patient reported outcome measure to assess physical function status. The scores range from 23.9 to 58. Higher the score, higher is the physical function.

SECONDARY OUTCOMES:
Average of all scores across the 6-items of Self-Efficacy for Managing Chronic Disease 6-Item (SEMCD-6) Scale | Baseline, Month 3, Month 6
  Scoring for each item is on a 1-10 scale where 1 is 'Not at all confident' and 10 is 'Totally Confident.' There are 6 such items. The scores of all the 6 items are combined and averaged to get the total score. The final score is between 1-10. Higher scores indicate higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Flores, PT, MSPT, MA, PhD, CLT, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States